CLINICAL TRIAL: NCT06298747
Title: Evaluation of the Efficacy of Ultrasound-guided Selective Cervical Root Pulsed Radiofrequency Therapy in Patients With Cervical Radicular Pain: Analysis of Single-Center Data
Brief Title: Ultrasound-guided Selective Cervical Root Pulsed Radiofrequency Therapy in Patients With Cervical Radicular Pain
Acronym: pulsedrf
Status: Completed | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Principal investigator, Diskapi Teaching and Research Hospital
Other Study IDs: Cervical root PRF
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Cervical Pain
Keywords: cervical radicular pain; ultrasonography; cervical nerve root; pulsed radiofrequency; analgesia
MeSH Terms: conditions — Neck Pain; Agnosia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Selective cervical nerve root pulsed radiofrequency: A 5-12 MHz linear US probe was used during the procedure. C7 has a more prominent posterior tubercle and a rudimentary anterior tubercle. C5 and C6 have more prominent and smooth anterior and posterior tubercles, respectively. After visualizing the hypoechoic nerve root between the tubercles of the transverse process, the surrounding vascular structures were identified and RF canula is used. After approaching the hypoechoic nerve root, after sensory and motor stimulation, PRF was applied to each nerve root with a current of 1.0-1.2 V at a frequency of 2 Hz for 4 minutes at 42 °C.
  Interventions: Other: Selective cervical nerve root pulsed radiofrequency

INTERVENTIONS:
Other: Selective cervical nerve root pulsed radiofrequency — A 5-12 MHz linear US probe was used during the procedure. C7 has a more prominent posterior tubercle and a rudimentary anterior tubercle. C5 and C6 have more prominent and smooth anterior and posterior tubercles, respectively. After visualizing the hypoechoic nerve root between the tubercles of the transverse process, the surrounding vascular structures were identified and RF canula is used. After approaching the hypoechoic nerve root, after sensory and motor stimulation, PRF was applied to each nerve root.

SUMMARY:
Chronic cervical pain is a common disorder with a prevalence of approximately 35% in adults. Cervical radicular pain is defined as radiating pain in the upper limb caused by compression or inflammation of the nerve roots ascending from the intervertebral foramen to the spinal cord, due to disc herniation or spinal stenosis. C7 and C6 are the two most commonly affected nerve roots. Various treatment modalities are available, including oral medications, physiotherapy, and epidural steroid injections. However, chronic and persistent pain that develops as a result of some patients not responding to these treatments. Ultrasound-guided selective cervical nerve root block and pulsed radiofrequency are interventional treatments used in patients with radicular cervical pain unresponsive to conservative treatments. Pulsed radiofrequency (PRF) treatment of peripheral nerves may provide long-term pain relief in patients with short-term pain relief with a local anesthetic block. Studies have shown the effectiveness of PRF therapy applied to selective cervical nerve roots in relieving cervical radicular pain.

DETAILED DESCRIPTION:
Pulsed radiofrequency treatment applied to selective cervical nerve roots (C5, C6, and C7) under ultrasound guidance is frequently used in patients with cervical radicular pain due to cervical disc herniation who do not respond adequately to medical treatment and physiotherapy.

Pain intensity was evaluated at baseline and 1,3 and 6 months after US-guided selective cervical nerve root PRF treatment using VAS (Visual analog scale). The primary outcome measure was percent reduction in pain, with 50% pain relief lasting at least 6 months was defined as a positive categorical outcome.

Patients' functionality and neuropathic pain status were assessed using the Neck Disability Index (NDI) and Douleur Neuropathique 4 Questions (DN4) at baseline and 1,3 and 6 months after US-guided selective cervical nerve root PRF treatment, respectively. Secondary outcome measure was defined as a positive categorical outcome of 50% or more improvement in these scores for at least 6 months.

In addition, demographic data such as age (years), gender, duration of pain (months), pain side (right or left), affected cervical nerve root level (one or multiple levels), and history of surgery for cervical disc herniation and analgesic use (nonsteroidal anti-inflammatory drugs or opioids) were obtained from patient data and retrospectively analyzed the patient's electronic medical history records.

The primary aim of this study was to determine the efficacy of US-SCNR PRF treatment, and the clinical and demographic variables associated with treatment outcomes. The secondary aim of this study was to determine the improvement in functionality and neuropathic pain status of patients after the procedure, and treatment-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* radicular pain radiating only to the neck and one arm for more than 12 weeks
* no response to conservative treatment (including analgesics and physiotherapy modalities)
* access to clinical data

Exclusion Criteria:

* inadequate medical records with missing Numerical Rating Scale (NRS), Neck Disability Index (NDI), and DN4 (Douleur Neuropathique 4 Questions) scores
* patients lost to follow-up within six months after the procedure
* history of malignancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with cervical radicular pain unresponsive to conservative treatments
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-02 (Actual)

PRIMARY OUTCOMES:
VAS | Change from Baseline VAS at 6 months
  Visual analogue scales (VAS) are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid (statistically measurable and reproducible) classification of symptom severity and disease control. (minimum value is 0 and maximum value is 10)

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | Change from Baseline NDI at 6 months
  NDI is a self-report questionnaire that measures the impact of neck pain on patient's daily activities and quality of life. It consists of ten items assessing pain intensity, self-care, lifting, reading, headache, concentration, work, driving, sleep, and leisure. Each item is scored between 0 and 5, with higher scores indicating more disability.
Douleur Neuropathique 4 Questions (DN4) | Change from Baseline NDI at 6 months
  The DN4 scale provides information on whether pain has a neuropathic character. It is scored according to the presence of burning, coldness, or electric shock sensation in the pain, tingling, numbness, stinging, or itching sensation in the same region, presence of touch or needle hypoesthesia on examination, and occurrence of pain in the same region with a brush. Although the maximum score was 10, a score >4 indicated the presence of neuropathic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Taylan Akkaya, MD, Study Director — Diskapi Teaching and Research Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided